CLINICAL TRIAL: NCT00087893
Title: Epidemiology of Vascular Inflammation & Atherosclerosis
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Russell Tracy, Professor of Pathology, University of Vermont
Other Study IDs: 1261; R01HL077449 (NIH)
Record Dates: First submitted 2004-07-15; First posted 2004-07-19 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Coronary Arteriosclerosis; Coronary Disease; Cerebral Arteriosclerosis; Cerebrovascular Accident
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Coronary Artery Disease; Coronary Disease; Intracranial Arteriosclerosis; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
To investigate the relationship of vascular cell phenotypes to atherosclerosis.

DETAILED DESCRIPTION:
BACKGROUND:

Currently, the predominant hypothesis regarding atherosclerosis is that it is in major part driven by two independent pathways: hyperlipidemia (the "stimulation") and inflammation (the "response"). Although vascular cells mediate the influence of inflammation on atherosclerosis, very little is known about vascular cell epidemiology and the relationship of vascular cell phenotypes to atherosclerosis. The main hypothesis tested in this study is that variation in vascular cell biology is related to the population variation in atherosclerosis.

DESIGN NARRATIVE:

The cross-sectional study will be nested within a large cohort study, the Multiethnic Study of Atherosclerosis (MESA). A partial sample of 1,000 individuals who have undergone other special laboratory analyses will be identified and new measures collected as part of their upcoming site visit. A number of novel cellular phenotypes describing the innate immune response (monocyte activation, natural killer and T cell counts), the adaptive immune response (TH1 and TH2 helper cells, and memory T cells), and vessel integrity (circulating endothelial progenitor cells) will be measured in these participants. Plasma constituents will also be measured that relate to the cellular phenotypes. The overall goal is to test the hypothesis that these novel phenotypes are associated with subclinical atherosclerosis in the coronary and carotid arteries assessed by quantification of coronary calcification (CAC) and B-mode ultrasound (CIMT), in addition to the other subclinical measures available from the MESA cohort.

ELIGIBILITY:
No eligibility criteria

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1,000 men and women aged 45-84 years
Sampling Method: Probability Sample
Enrollment: 931 (Actual)
Dates: Start 2004-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
T helper bias | 2008
  T helper bias is a stable phenotype in people, with few environmental drives; the main environmental driver appears to be anti-CMV titer; this has led to our view that genetics probably plays a role, and our current GWAS efforts using our unique MESA-Inflammation cellular phenotypes.

SECONDARY OUTCOMES:
T helper bias toward Th1 cells | 2008
  T helper bias towards Th1 cells is strongly associated with measures of atherosclerosis in the population-based study MESA-Inflammation (both coronary calcification and carotid wall thickness) after fully adjusting for traditional and novel CVD risk factors. This is consistent with our original hypothesis, based on small human studies and mouse data.

OTHER OUTCOMES:
atherosclerosis | 2008
  Both IL-10 and sIL-2R are also associated with atherosclerosis in humans as we hypothesized.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Tracy, Principal Investigator — University of Vermont